CLINICAL TRIAL: NCT05878418
Title: The Effect of Spinal Orthosis on the Development of Scoliosis and Chest Deformity in Type I Spinal Muscular Atrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Emre DANSUK, MSc, Physiotherapist, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-772.02-200
Record Dates: First submitted 2023-05-09; First posted 2023-05-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Spinal Muscular Atrophy Type I; Scoliosis; Chest Deformities; Spinal Orthosis; Pulmonary Rehabilitation; Exercise
Keywords: Spinal Muscular Atrophy Type I; Scoliosis; Chest Deformities; Spinal Orthosis; Pulmonary Rehabilitation; Exercise
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood; Scoliosis; Motor Activity | interventions — Respiratory Therapy

STUDY DESIGN:
Intervention Model Description: Parallel Assignment randomised controlled trial
Who Masked: Participant
Masking Description: Participants will not know which group to belong to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trunk Exercises, Pulmonary Rehabilitation and Pulmonary Care Program + Spinal Orthosis Group (Experimental): Trunk Exercises, Pulmonary Rehabilitation and Pulmonary Care Program + Toracolumbosacral Spinal Orthosis
  Interventions: Device: Thoracolumbosacral Spinal Orthosis (TLSO); Other: Trunk Exercise (TE), Pulmonary Rehabilitation(PR) and Pulmonary Care (PC)
- Trunk Exercises, Pulmonary Rehabilitation and Pulmonary Care Program Group (Active Comparator): Trunk Exercises, Pulmonary Rehabilitation and Pulmonary Care Program
  Interventions: Other: Trunk Exercise (TE), Pulmonary Rehabilitation(PR) and Pulmonary Care (PC)

INTERVENTIONS:
Device: Thoracolumbosacral Spinal Orthosis (TLSO) — In the TE, PR, PC + spinal orthosis group, in addition to the control group program, a thoracolumbosacral spinal orthosis (TLSO) designed specifically for the child will be used for 8 hours a day for 8 weeks, every day of the week.
  Other Names: Pulmonary Rehabilitation; Pulmonary Care; Trunk Exercise
  Arms: Trunk Exercises, Pulmonary Rehabilitation and Pulmonary Care Program + Spinal Orthosis Group
Other: Trunk Exercise (TE), Pulmonary Rehabilitation(PR) and Pulmonary Care (PC) — The active control group will receive a TE, PR and PC program in the outpatient clinic once a week for 8 weeks, 7 days a week, once a day, 50-60 minutes per session, for 8 weeks.

SUMMARY:
Spinal muscular atrophy (SMA) is a serious neuromuscular disease characterized by the degeneration of alpha motor neurons in the spinal cord, resulting in progressive proximal muscle atrophy and denervation. The main problems are posture disorders, scoliosis, pelvic curvature, contracture, hip dislocation, foot and chest deformities. In this study, examining the effectiveness of trunk support used to alleviate the progression of scoliosis in children diagnosed with SMA Type I will contribute to the current literature.In addition to Individualized Trunk Exercises (ITE), Individualized Pulmonary Rehabilitation (IPR) and Chest Care (CC) Programme, the use of thoracolumbosacral spinal orthosis in Type I children will be used for the first time in our country and in the world literature. SMA. Our aim in the project is to examine the effectiveness of this treatment program on the motor functions, scoliosis Cobb angle, pelvic curvature and chest deformity of children with Type I SMA.The project is planned to be carried out with children diagnosed with Type I SMA who are followed up at Medipol Mega University Hospital Pediatric Chest Diseases Polyclinic.In evaluating the development of scoliosis as the primary outcome measure; Radiological evaluation (Cobb Angle) and examination of chest deformity; Lung X-ray (Basal Chest Wall Upper-Lower Ratio Measurement) will be used. As secondary outcome measures, the Children's Hospital of Philadelphia Infant Test for Neuromuscular Disorders and the Hammersmith Functional Motor Scale Expanded were used to assess motor functions and examine the level of motor development; In the World Health Organization Motor Development Scale body posture assessment; Supine Trunk Rotation Angle Test and Pelvic Curvature Test, pulse oximetry to assess oxygenation; In determining the level of satisfaction with orthosis use; Children/families' information will be questioned through the Quebec Assistive Technology User Satisfaction Evaluation Survey and Personal Information Form.The active control group will receive the ITE, IPR and CC program as a home program and once a week in the outpatient clinic for 8 weeks, 7 days a week, once a day, each session being 50-60 minutes. In the ITE-IPR-CC + spine orthosis group, in addition to the control group program, a thoracolumbosacral spine orthosis specially designed for the child will be used every day of the week and 8 hours a day for 8 weeks. Evaluations will be made at baseline and at week 8.

DETAILED DESCRIPTION:
With the increase in scoliosis and scoliosis-related symptoms after increased survival in patients with Type I SMA, the need for physiotherapy applications has become more important than ever (Trenkle, et al., 2021; Mercuri, et al., 2018). The presence of scoliosis significantly affects lung capacity, postural control, functionality and quality of life in patients with Type I SMA. For this reason, it is of great importance to treat these patients in a timely and effective manner. There is no consensus on the type of spinal orthosis and application protocol to be used in patients with SMA (Mercuri, et al., 2018). When the literature was examined, no study was found about the effect of spinal orthosis use on scoliosis and chest deformity in Type I SMA patients.

ELIGIBILITY:
Inclusion Criteria:

* 2-6 years old,
* Clinically and genetically diagnosed as Type I SMA,
* Having scoliosis (20-40 Cobb angle),
* Children who have not had any previous spinal surgery,
* Children who have received or continue to receive their medical treatments (nusinersen and onasemnogene abeparvovec).

Exclusion Criteria:

* Having acute respiratory failure and/or serious airway infections,
* 24-hour mechanical ventilation dependency,
* Continuing medical treatment in intensive care,
* Having other orthopedic and neurological problems,
* Children of parents who did not agree to participate in the study,
* Children whose chest expansion and/or oxygenation are at risk of being affected and who cannot tolerate the orthosis,
* Children and their parents who do not use the thoracolumbosacral spinal orthosis in accordance with the study protocol and do not comply with trunk exercises, pulmonary rehabilitation and pulmonary care practices.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-10-11 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Radiological Evaluation (Cobb Angle) | 8 week
  The presence of scoliosis will initially be evaluated clinically using spinal x-rays. The Cobb angle will be used as a measure of scoliosis progression. If possible, radiological evaluation will be performed in the assisted sitting position without providing sitting balance, if it is difficult to take X-rays in the sitting position, in the supine position. Two images will be obtained, anteroposterior and lateral. The location of scoliosis will be classified as thoracic, thoracolumbar and lumbar. Scoliosis direction will be recorded as right and left. In the case of S-shaped scoliosis, the angle used for assessment will be the highest degree.
Lung X-ray (Basal Chest Wall Upper-Lower Ratio Measurement) | 8 week
  The anteroposterior view of the chest radiograph taken in the supine position will be used. A perpendicular line will be drawn connecting the spinous processes to the horizontal lines drawn from the inner edge of the rib. The longest line of the 2nd rib (Dapex(upper)) and the 9th rib (Dbase(lower)) will be measured. The percentage ratio of the upper/lower chest wall will be calculated as Dapex(upper) / Dbase(lower)×100(%). The presence of pulmonary problems such as atelectic areas will be determined on the chest radiograph and the change in trunk diameter and depth during thoracic expansion will be monitored.

SECONDARY OUTCOMES:
Philadelphia Children's Hospital Infant Test of Neuromuscular Disorders (CHOP-INTEND) | 8 week
  Philadelphia Children's Hospital Infant Test for Neuromuscular Disorders (CHOP-INTEND) will be used to evaluate motor functions. The CHOP INTEND is a functional scale that has been shown to reliably assess motor function in patients with infancy-onset Type I SMA and other neuromuscular disorders. The development of the scale is based on the natural history of motor function progression for infants with Type I SMA. The test contains 16 items that provide information on muscle strength and function, gravity eliminated, gravity assisted, and antigravity. Items are ranked from easy to difficult, with the least tolerated items being tested last.
  * Scoring: rated from 0 (no response) to 4 (complete response). The maximum score is 64.
  * Application time: It can be completed in 15-40 minutes.
  * Equipment: mat, rattle, plush toy, toy phone.
Hammersmith Extended Functional Motor Scale (HFMSE) | 8 week
  Hammersmith Functional Motor Scale Extended Version (HFMSE) will be used to evaluate motor functions. The HFMSE test consists of 33 items in which movements such as sitting, rolling in the supine position, raising the head in the lying position, standing up, kneeling, standing and stepping, jumping, and climbing stairs are scored. Each item is evaluated on a scoring system with 2 points for "can do without support", 1 point for "can do with support" and 0 points for "can't".
  The scores of all items are summed, the total score ranges from 0 to 66, and a higher score means better motor functions.
World Health Organization Motor Development Scale (WHO Developmental Milestones) | 8 week
  With the World Health Organization Motor Development Scale, 6 different gross motor levels will be evaluated as unsupported sitting, hand-knee crawling, assisted standing, assisted walking, standing alone and walking alone.
Supine Trunk Rotation Angle Test | 8 week
  Chest deformity will be measured using a scoliometer (Basic Economics). The patient will be in the supine position with the head symmetrical. Scoliometer, 2nd-3rd in the upper part of the sternum. it will be located along the chest at the level of the rib (SATR upper) and below the sternum, where the corpus meets the xiphoid process of the sternum (SATR lower).
Pelvic Tilt Test | 8 week
  Pelvic tilt measurement will be made using a scoliometer (Basic Economics) placed at the posterior superior iliac spines in a modified sitting position with supported upper and lower extremities.
Quebec Assistive Technology User Satisfaction Assessment Questionnaire (QUEST) | 8 week
  The Quebec Assistive Technology User Satisfaction Assessment Questionnaire (QUEST) will be used to assess spinal orthosis satisfaction. Since the patients are in childhood, the questionnaire will be filled in by their parents. Interviews will be conducted face to face. Responses are scored on a 5-point Likert scale for satisfaction (1=very dissatisfied and 5=very satisfied). The QUEST questionnaire has 3 points; these are device satisfaction, service satisfaction and total score. Satisfaction defined in the questionnaire is the individual's critical evaluation of the technological device. The individual's expectations, perception, attitude and personal characteristics affect this evaluation. The QUEST questionnaire contains 12 items questioning the satisfaction of the assistive device (8 items) and the service (4 items). At the end of the questionnaire, individuals/parents are asked to select and mark 3 of the 12 items as important.
Respiratory Evaluation | 8 week
  Respiratory type, frequency and oxygen saturation will be examined. Respiratory type; It will be determined whether the patient has thoracic, abdominal, thoracoabdominal breathing or pursed-lip breathing. Respiratory frequency; It will be recorded as the number of respirations taken and exhaled per minute. Although the normal respiratory frequency is 12-20 respiratory rates/minute; <12 respiratory rate/minute is called bradypnea, >12 respiratory rate/minute is called tachypnea. Oxygen saturation measurement will be carried out by attaching the Contec brand CMS60D handheld pulse oximeter device, which is available at our university, to the children's toes before wearing the corset, while the corset is put on and 10 minutes after the corset is put on.

OTHER OUTCOMES:
Personal Information Form | Baseline
  With the personal information form, the age, gender, weight, height, type of diagnosis, age of diagnosis, type of delivery, auxiliary equipment (orthotics, body support, mobility aids; wheelchair, walker, etc.) and drug use of the patients will be recorded. The age, education level, marital status, number of births, economic status, social security and number of people living in the household will also be noted.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Dansuk, MSc, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dansuk E, Van Den Berg ANT, Ata G, Yikilmaz SK, Oktem S. The effect of thoracolumbosacral orthosis on scoliosis progression and chest deformity in children with type 1 spinal muscular atrophy: A randomized controlled trial. PLoS One. 2025 Sep 15;20(9):e0323341. doi: 10.1371/journal.pone.0323341. eCollection 2025. PMID 40953000